CLINICAL TRIAL: NCT06817746
Title: Fostering Infant Responsivity and Reciprocity - Support to Thrive. A Multisite Randomized Control Trial of a Preemptive Telehealth Intervention for Infants With Early Signs of Autism Spectrum Disorders
Brief Title: Telehealth Intervention for Infants With Prodromes of ASD
Acronym: FIRRST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Policlinico Hospital/University of Messina (Unknown); CNR Messina (Unknown); Istituto Italiano di Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FIRRST_VIITA
Record Dates: First submitted 2025-01-21; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Autism Spectrum Disorder (ASD); ASD Prodromes; Infants; Support; Pre-emptive; Parent Mediated
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FIRRST (Experimental): FIRRST is based on the principles of Naturalistic Developmental Behavioral Interventions (NDBIs), and more specifically on the principles of Infant Start and iBASIS. FIRRST targets ASD prodromes including diminished eye contact, diminished communicative intent, diminished social orientation, and unusual pattern of object exploration. Additionally, it also targets motor immaturity, frequent in infants at risk for ASD. FIRRST is a systemic approach, integrated within the family dynamics and culture. The program will address the five elements identified in efficacious very early intervention: 1) parent involvement, 2) frequency and length of intervention, 3) individualized, developmentally appropriate activities, 4) beginning the interventions as early as possible, and 5) increasing parental sensitivity and responsivity to infant cues. FIRRST will be delivered by experienced licensed health professionals trained by the developer of the intervention.
  Interventions: Behavioral: FIRRST
- Parent Education (Active Comparator): Families will receive written educational material focused on supporting child development and targeting ASD specific immaturities and atypicalities. Additionally, parent education families will receive counseling once per month for 6 months delivered by a licensed health professional aiming at supporting the family well being and helping the family to connect with the local public health services.
  Interventions: Behavioral: Parent Education

INTERVENTIONS:
Behavioral: FIRRST — FIRRST is based on the principles of Naturalistic Developmental Behavioral Interventions (NDBIs), and more specifically on the principles of Infant Start and iBASIS. FIRRST targets ASD prodromes including diminished eye contact, diminished communicative intent, diminished social orientation, and unusual pattern of object exploration. Additionally, it also targets motor immaturity, frequent in infants at risk for ASD. FIRRST is a systemic approach, integrated within the family dynamics and culture. The program will address the five elements identified in efficacious very early intervention: 1) parent involvement, 2) frequency and length of intervention, 3) individualized, developmentally appropriate activities, 4) beginning the interventions as early as possible, and 5) increasing parental sensitivity and responsivity to infant cues. FIRRST will be delivered by experienced licensed health professionals trained by the developer of the intervention.
  Arms: FIRRST
Behavioral: Parent Education — Families will receive written educational material focused on supporting child development and targeting ASD specific immaturities and atypicalities. Additionally, parent education families will receive counseling once per month for 6 months delivered by a licensed health professional aiming at supporting the family well being and helping the family to connect with the local public health services.
  Arms: Parent Education

SUMMARY:
Autism Spectrum Disorder (ASD) is a complex neurodevelopmental disorder characterized by social-communication and interaction deficits and restricted, repetitive patterns of interests and behavior. It is frequently associated with heterogeneous comorbidities including physical, mental, and neurodevelopmental disorders, which can result in a substantial burden on individuals, families, and society.

Early prodromal signs of ASD emerge during the first year of life, a time when brain plasticity is at its maximum level, and may consist of diminished social orienting, responsivity and reciprocity combined with the presence of prolonged visual fixation and repetitive use of objects. Developmental immaturities in communication and motor skills are often present too. Pre-emptive Intervention (PI) for infants with prodromal signs of ASD was shown to improve outcomes, in comparison to later starts, by improving developmental skills, reducing ASD symptoms and, in some cases, preventing the full blown symptoms of ASD. Moreover, access to early evidence-based interventions may reduce the elevated levels of stress, anxiety and depressive symptoms experienced by caregivers of children with signs of ASD.

Despite this evidence, professionals tend to have a 'wait to see' approach, rather than targeting areas of impairment with early intervention. Moreover, the vast majority of current clinical models of ASD services require a diagnosis to receive services, while the identification of prodromal signs of the disorders generally is not sufficient to access early intervention. There is an urgent need for a paradigm shift in ASD treatment.

The proposed Project aims to evaluate the efficacy of FIRRST, a parent-mediated PI for infants with early signs of ASD. We will conduct a multisite RCT of telehealth PI by recruiting 132 symptomatic infants between 9-14 months and randomly assigning them to receive either FIRSST (experimental group), or Parent Education (control group). Developmental skills, ASD symptomatology, caregiver well-being and brain changes on High-Density EEG will be assessed with in-presence evaluations at three time points: 1. baseline; 2. after 24 weeks of intervention; 3. follow-up after 24 weeks from the end of intervention.

If funded, The proposed study will be the first well-powered RCT evaluating developmental, symptom and neurophysiological changes in response to a parent-mediated PI conducted in Europe. The ultimate goal for translational research in ASD lies in the optimization of clinical outcomes through the most effective, targeted, and timely treatments. The proposed RCT has the potential to significantly impact current access to services by reducing the age of starting intervention, thereby promoting optimal developmental outcomes, as well as reducing burden and high health costs to families and society.

ELIGIBILITY:
Inclusion Criteria:

* risk-range score at SACS-R;
* Italian as one of the languages spoken at home;
* age below 18 months (corrected) at the time of identification;
* available device with webcam and home internet access.

Exclusion criteria:

* presence of a known genetic disorder, brain damage or other relevant neurological or chronic disorders;
* severe visual, auditory and/or motor impairment.

Ages: 9 Months to 17 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Infant Development | T0: at recruitment; T1: after 6 months since recruitment; T2: after 12 months since recruitment.
  The Griffiths III, a scale to assess developmental quotients (Green et al., 2016).
ASD Symptom Severity | T0: at recruitment; T1: after 6 months since recruitment; T2: after 12 months since recruitment.
  The Autism Diagnostic Observation Schedule-Second Edition (ADOS-2) Toddler Module, to assess clinical severity of autism (Lord et al., 2012)
Change of Core ASD Symptoms | T0: at recruitment; T1: after 6 months since recruitment; T2: after 12 months since recruitment.
  The Brief Observation of Social Communication Change (BOSCC) to measure change of core ASD symptoms (Gradzinski et al., 2016) in response to intervention.

SECONDARY OUTCOMES:
Parent Mental Well-Being | T0: at recruitment: T1: after 6 months since recruitment; T2: after 12 months since recruitment.
  The Parenting Stress Index-4 (PSI-4), to evaluate the magnitude of stress in the parent-child system (Abidin, 2016).
Parent-Child Interaction | T0: at recruitment; T1: after 6 months since recruitment; after 12 months since recruitment.
  The MONSI-CC (Measure of NDBI Strategy Implementation-Caregiver Change) to evaluate changes in parent-child interaction style in response to intervention.
Neurophysiological Modifications | To: at recruitment; T1: after 6 months since recruitment; T2: after 12 months since recruitment.
  Modifications in HD-EEG activity in terms of 1/f aperiodic signal.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Guzzetta, MD, Principal Investigator — University of Pisa/IRCCS Stella Maris; Sara Calderoni, MD, Principal Investigator — University of Pisa/IRCCS Stella Maris; Costanza Colombi, PhD, Principal Investigator — IRCCS Stella Maris; Lilian Ruta, MD, Principal Investigator — CNR Messina; Gabriella Di Rosa, MD, Principal Investigator — University of Messina; Michale Lombardo, PhD, Principal Investigator — Istituto Italiano Tecnologia
Locations (4):
- Italy (4):
  - IRCCS Stella Maris, Pisa, Italy
  - Istituto Italiano Tecnologia, Rovereto, Italy
  - CNR, Messina
  - University of Messina, Messina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xiao Y, Wen TH, Kupis L, Eyler LT, Taluja V, Troxel J, Goel D, Lombardo MV, Pierce K, Courchesne E. Atypical functional connectivity of temporal cortex with precuneus and visual regions may be an early-age signature of ASD. Mol Autism. 2023 Mar 10;14(1):11. doi: 10.1186/s13229-023-00543-8. PMID 36899425
- [Background] Bertelsen N, Landi I, Bethlehem RAI, Seidlitz J, Busuoli EM, Mandelli V, Satta E, Trakoshis S, Auyeung B, Kundu P, Loth E, Dumas G, Baumeister S, Beckmann CF, Bolte S, Bourgeron T, Charman T, Durston S, Ecker C, Holt RJ, Johnson MH, Jones EJH, Mason L, Meyer-Lindenberg A, Moessnang C, Oldehinkel M, Persico AM, Tillmann J, Williams SCR, Spooren W, Murphy DGM, Buitelaar JK; EU-AIMS LEAP group; Baron-Cohen S, Lai MC, Lombardo MV. Imbalanced social-communicative and restricted repetitive behavior subtypes of autism spectrum disorder exhibit different neural circuitry. Commun Biol. 2021 May 14;4(1):574. doi: 10.1038/s42003-021-02015-2. PMID 33990680
- [Background] Loth E, Charman T, Mason L, Tillmann J, Jones EJH, Wooldridge C, Ahmad J, Auyeung B, Brogna C, Ambrosino S, Banaschewski T, Baron-Cohen S, Baumeister S, Beckmann C, Brammer M, Brandeis D, Bolte S, Bourgeron T, Bours C, de Bruijn Y, Chakrabarti B, Crawley D, Cornelissen I, Acqua FD, Dumas G, Durston S, Ecker C, Faulkner J, Frouin V, Garces P, Goyard D, Hayward H, Ham LM, Hipp J, Holt RJ, Johnson MH, Isaksson J, Kundu P, Lai MC, D'ardhuy XL, Lombardo MV, Lythgoe DJ, Mandl R, Meyer-Lindenberg A, Moessnang C, Mueller N, O'Dwyer L, Oldehinkel M, Oranje B, Pandina G, Persico AM, Ruigrok ANV, Ruggeri B, Sabet J, Sacco R, Caceres ASJ, Simonoff E, Toro R, Tost H, Waldman J, Williams SCR, Zwiers MP, Spooren W, Murphy DGM, Buitelaar JK. The EU-AIMS Longitudinal European Autism Project (LEAP): design and methodologies to identify and validate stratification biomarkers for autism spectrum disorders. Mol Autism. 2017 Jun 23;8:24. doi: 10.1186/s13229-017-0146-8. eCollection 2017. PMID 28649312
- [Background] Garces P, Baumeister S, Mason L, Chatham CH, Holiga S, Dukart J, Jones EJH, Banaschewski T, Baron-Cohen S, Bolte S, Buitelaar JK, Durston S, Oranje B, Persico AM, Beckmann CF, Bougeron T, Dell'Acqua F, Ecker C, Moessnang C, Charman T, Tillmann J, Murphy DGM, Johnson M, Loth E, Brandeis D, Hipp JF; EU-AIMS LEAP group authorship. Resting state EEG power spectrum and functional connectivity in autism: a cross-sectional analysis. Mol Autism. 2022 May 18;13(1):22. doi: 10.1186/s13229-022-00500-x. PMID 35585637
- [Background] Santocchi E, Guiducci L, Fulceri F, Billeci L, Buzzigoli E, Apicella F, Calderoni S, Grossi E, Morales MA, Muratori F. Gut to brain interaction in Autism Spectrum Disorders: a randomized controlled trial on the role of probiotics on clinical, biochemical and neurophysiological parameters. BMC Psychiatry. 2016 Jun 4;16:183. doi: 10.1186/s12888-016-0887-5. PMID 27260271
- [Background] Aiello S, Leonardi E, Cerasa A, Servidio R, Fama FI, Carrozza C, Campisi A, Marino F, Scifo R, Baieli S, Corpina F, Tartarisco G, Vagni D, Pioggia G, Ruta L. Video-Feedback Approach Improves Parental Compliance to Early Behavioral Interventions in Children with Autism Spectrum Disorders during the COVID-19 Pandemic: A Pilot Investigation. Children (Basel). 2022 Nov 8;9(11):1710. doi: 10.3390/children9111710. PMID 36360438
- [Background] Whitehouse AJO, Varcin KJ, Pillar S, Billingham W, Alvares GA, Barbaro J, Bent CA, Blenkley D, Boutrus M, Chee A, Chetcuti L, Clark A, Davidson E, Dimov S, Dissanayake C, Doyle J, Grant M, Green CC, Harrap M, Iacono T, Matys L, Maybery M, Pope DF, Renton M, Rowbottam C, Sadka N, Segal L, Slonims V, Smith J, Taylor C, Wakeling S, Wan MW, Wray J, Cooper MN, Green J, Hudry K. Effect of Preemptive Intervention on Developmental Outcomes Among Infants Showing Early Signs of Autism: A Randomized Clinical Trial of Outcomes to Diagnosis. JAMA Pediatr. 2021 Nov 1;175(11):e213298. doi: 10.1001/jamapediatrics.2021.3298. Epub 2021 Nov 1. PMID 34542577
- [Background] Rogers SJ, Vismara L, Wagner AL, McCormick C, Young G, Ozonoff S. Autism treatment in the first year of life: a pilot study of infant start, a parent-implemented intervention for symptomatic infants. J Autism Dev Disord. 2014 Dec;44(12):2981-95. doi: 10.1007/s10803-014-2202-y. PMID 25212413
- [Background] Lombardo MV, Busuoli EM, Schreibman L, Stahmer AC, Pramparo T, Landi I, Mandelli V, Bertelsen N, Barnes CC, Gazestani V, Lopez L, Bacon EC, Courchesne E, Pierce K. Pre-treatment clinical and gene expression patterns predict developmental change in early intervention in autism. Mol Psychiatry. 2021 Dec;26(12):7641-7651. doi: 10.1038/s41380-021-01239-2. Epub 2021 Aug 2. PMID 34341515
- [Background] Bosl WJ, Tager-Flusberg H, Nelson CA. EEG Analytics for Early Detection of Autism Spectrum Disorder: A data-driven approach. Sci Rep. 2018 May 1;8(1):6828. doi: 10.1038/s41598-018-24318-x. PMID 29717196
- [Background] Jones W, Klin A. Attention to eyes is present but in decline in 2-6-month-old infants later diagnosed with autism. Nature. 2013 Dec 19;504(7480):427-31. doi: 10.1038/nature12715. Epub 2013 Nov 6. PMID 24196715
- See also: Related Info — https://www.fsm.unipi.it
- Available data/document: Study Protocol — https://www.fsm.unipi.it